CLINICAL TRIAL: NCT07252284
Title: China Adrenal Venous Sampling Investigation: A National Multicenter Study
Brief Title: CHina Adrenal Venous saMPling InvestigatiON
Acronym: CHAMPION
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Hui DONG, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2024-2484
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hyperaldosteronism; Adrenal Venous Sampling; Adrenalectomy
Keywords: Adrenal venous sampling; Hyperaldosteronism; Antecubital approach; Femoral approach; Main adverse cardiovascular events
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adrenal Venous Sampling: Patients with Primary Aldosteronism (PA) undergoing Adrenal Venous Sampling via antecubital approach or femoral approach to discriminate PA forms with unilateral from bilateral excess aldosterone production.
  Interventions: Procedure: adrenal venous sampling

INTERVENTIONS:
Procedure: adrenal venous sampling — Patients with Primary Aldosteronism (PA) undergoing Adrenal Venous Sampling via antecubital approach or femoral approach to discriminate PA forms with unilateral from bilateral excess aldosterone production.

SUMMARY:
Primary aldosteronism (PA) is a major cause of secondary hypertension, yet its optimal diagnosis and management remain challenging. This study comprehensively evaluates adrenal venous sampling (AVS), addressing key clinical, technical, and methodological issues, and aims to clarify the relationship between AVS-guided management and long-term clinical and biochemical outcomes to optimize patient care and prognosis.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is one of the most common causes of secondary hypertension, yet its optimal diagnostic and therapeutic strategies remain challenging. Adrenal venous sampling (AVS) is regarded as the gold standard for subtype differentiation; however, important clinical, technical, and methodological issues have not been systematically addressed. This study is designed to comprehensively evaluate AVS and its clinical implications, aiming to elucidate the relationship between AVS-guided diagnosis and management of PA and long-term clinical and biochemical outcomes, while refining AVS protocols, standardizing clinical practice, optimizing therapeutic decision-making, and ultimately improving patient management and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed primary aldosteronism;
2. Patients undergoing adrenal venous sampling for subtype classification of primary aldosteronism.

Exclusion Criteria:

1. Severe comorbidity, including stroke, myocardial infarction, heart failure, severe valvular heart disease, liver cirrhosis, and metastatic tumor within the previous 3 months；
2. An estimated glomerular filtration rate <45 ml/min/1.73 m2, or serum creatinine >176 μmol/L；
3. Patients who refuse adrenalectomy;
4. Suspected of having an adrenocortical carcinoma;
5. Allergy to contrast agent;
6. Pregnant, nursing, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with confirmed primary aldosteronism underwent adrenal venous sampling.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) at 1-year follow-up | 1 year after AVS procedure
  Incidence of major adverse cardiovascular events (MACE) at 1-year follow-up, including stroke, heart failure, severe arrhythmias, renal failure, myocardial infarction, and death.

SECONDARY OUTCOMES:
The success rate of left adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)
The success rate of right adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)
The success rate of bilateral adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)
Selection of intraoperative catheter | At AVS procedure
  Types of catheter at the time of Adrenal Venous Sampling via antecubital approach or femoral approach
Time of the procedure | At AVS procedure
  Time of the procedure
Time of fluoroscopy | At AVS procedure
  Time of fluoroscopy
The contrast agent dosage | At AVS procedure
  The contrast agent dosage
the incidence of complications | 1 week after AVS procedure
  Complications related to adrenal vein cannulations (adrenal vein hematoma, inferior vena cava dissection, puncture site hematoma, etc)
the cost of the procedure | At AVS procedure
  the cost of the procedure
Change in 24-hour ambulatory systolic blood pressure | At 1, 3, 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after treatment
  The difference in average systolic blood pressure measured by 24-hour ambulatory blood pressure monitoring (ABPM) between baseline and each follow-up time point.
Change in 24-hour ambulatory diastolic blood pressure | At 1, 3, 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after treatment
  The difference in average diastolic blood pressure measured by 24-hour ambulatory blood pressure monitoring (ABPM) bewteen baseline and each follow-up time point.
Change in office systolic blood pressure | At 1, 3, 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after treatment
  The difference in systolic blood pressure measured during clinic visits (office blood pressure) between baseline and each follow-up time point
Change in office diastolic blood pressure | At 1, 3, 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after treatment
  The difference in diastolic blood pressure measured during clinic visits (office blood pressure) between baseline and each follow-up time point
Change in antihypertensive medication burden | At 1, 3, 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after treatment
  The change in the number and/or dosage of antihypertensive medications taken by patients between baseline and each follow-up time point
Change in urinary albumin-to-creatinine ratio (UACR) | At 1, 3, 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after treatment
  The difference in urinary albumin-to-creatinine ratio measured at baseline and at each follow-up time point
Change in left ventricular mass index (LVMI) | At 1, 3, 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after treatment
  The change in left ventricular mass index, as assessed by echocardiography, from baseline to each follow-up time point.
Change in pulse wave velocity (PWV) from baseline | At 1, 3, 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after treatment
  The change in pulse wave velocity measured between baseline and each follow-up time point。
Clinical Outcome According to Primary Aldosteronism Surgical Outcome (PASO) Criteria | At 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after surgery
  Clinical outcomes will be assessed at each follow-up visit afteradrenal surgery according to the PASO consensus criteria. Outcomes will be categorized as:
  (1)Complete clinical success: normal blood pressure without the need for any antihypertensive medication. (2)Partial clinical success: improvement in blood pressure and/or a reduction in the number or dosage of antihypertensive medications. (3)Absent clinical success: no improvement in blood pressure or antihypertensive medication burden.
Biochemical Outcome According to Primary Aldosteronism Surgical Outcome (PASO) Criteria | At 6, 12, and 18 months; and 2, 3, 4, 5, and 10 years after surgery
  Biochemical outcomes will be assessed at each follow-up visit after adrenal surgery according to the PASO consensus classification. Outcomes will be categorized as:(1)Complete biochemical success: normal serum potassium levels and a normalized aldosterone-to-renin ratio (ARR) without the need for potassium supplementation.(2)Partial biochemical success: improvement in biochemical parameters without full normalization.(3)Absent biochemical success: no improvement in biochemical markers compared to baseline.
Major adverse cardiovascular events (MACE) | At 6 and 18 months; and 2, 3, 4, 5, and 10 years after AVS procedure
  Incidence of major adverse cardiovascular events (MACE), including stroke, heart failure, severe arrhythmias, renal failure, myocardial infarction, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Dong, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (76):
- China (76):
  - The first affiliated hospital of USTC, Hefei, Anhui
  - Chuiyangliu Hospital affiliated to Tsinghua University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Central Hospital, Chongqing, Chongqing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - People's Hospital Affiliated to ChongqingThree Gorges Medical college, Chongqing, Chongqing Municipality
  - First Affiliated Hospital, Fujian Medical University, Fuzhou, China,, Fuzhou, Fujian
  - Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Forth People's Hosptal of Nanhai District of Foshan City, Foshan, Guangdong
  - Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Guangzhou, Guangdong
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, Guangdong
  - Shenzhen Third People's Hospital，Shenzhen, Guangdong Province 518112, China, Shenzhen, Guangdong
  - Shenzhen Dapeng New District Kuiyong People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Affliated Hospital Of GuangXi Medical Univesity, Nanning, Guangxi
  - Nanning Third People's Hospital, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou 550002, China., Guiyang, Guizhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Affiliated Hospital Of Guizhou Medical University, Kaili, Guizhou
  - Hainan General Hospital, Department of Endocrinology, Haikou, Hainan
  - Hainan General Hospital, Department of Cardiology, Hainan, Hainan
  - Tangshan hongci Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Kai Feng the Peoples Hospital, Kaifeng, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou Central Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou Yihe Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Affiliated Hospital of Hubei University of Arts and Science, Xiangyang, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Zhuzhou Hospital Affiliated to Xiangya School of Medicine,Central South University, Zhuzhou, Hunan
  - Xuzhou Central Hospital, Jiangsu, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Provincial People's Hospital (The First Affiliated Hospital of Nanchang Medical College), Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin Province FAW General Hospital, Changchun, Jilin
  - Affilated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Frist Aiffiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The second hospital of Dalian Medical University, Dalian, Liaoning
  - Inner Mongolia Xing'an League People's Hospital, Ulanhot, Neimenggu
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - Qinghai Province Cardiovascular and Cerebrovascular Disease Specialist Hospital, Xining, Qinghai
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - the Second Hospital, Cheeloo College of Medicine, Shandong University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - People's Hospital of Donga County, Shandong Province, Liaocheng, Shandong
  - Qingdao Hospital University of Health and Rehabilitation Sciences (Qingdao Municipal Hospital), Qingdao, Shandong
  - Shanghai Institute of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Putuo District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital ( originally named Shanghai First People's Hospital), Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - the second hospital of ShanXi medical unversity, Taiyuan, Shanxi
  - Xi'an People's Hospital, Xi’an, Shanxi
  - The Affiliated Hospital of Southwest Jiaotong University, The Third People's Hospital of Chengdu, Chengdu, China, Chengdu, Sichuan
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality
  - Changdu People's Hospital of Tibet, Chamdo, Tibet
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - Yili Kazak Autonomous Prefecture Friendship Hospital, Yining, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yan'an Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan
  - Zhejiang Hospital, Hangzhou, Zhejiang